CLINICAL TRIAL: NCT06396637
Title: The Efficacy and Safety of PD-1 Antibody Combined With Sapropterin Dihydrochloride in Patients With Advanced Pancreatic Cancer Who Failed to Standard Treatment.
Brief Title: PD-1 Antibody and Sapropterin Dihydrochloride in Patients With PDAC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Rui-hua Xu, MD, PhD, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-PDAC
Record Dates: First submitted 2024-04-30; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Adenocarcinoma Metastatic
Keywords: Pancreatic adenocarcinoma; PD-1 inhibitor
MeSH Terms: interventions — sapropterin; spartalizumab

STUDY DESIGN:
Intervention Model Description: PD-1 Antibody combined with Sapropterin Dihydrochloride
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): PD-1 Antibody combined with Sapropterin Dihydrochloride
  Interventions: Drug: Sapropterin Dihydrochloride

INTERVENTIONS:
Drug: Sapropterin Dihydrochloride — Sapropterin Dihydrochloride: 20mg/kg, qd
  Other Names: PD-1 Antibody

SUMMARY:
The prognosis for pancreatic cancer remains dismal, with current guidelines favoring FOLFIRINOX or AG (consisting of Gemcitabine and Abraxane) as the primary chemotherapeutic option. However, research has indicated limited benefits for patients with pancreatic cancer undergoing immunotherapy using Anti-PD-1 antibodies. In this context, researchers aim to investigate the therapeutic potential of Sapropterin Dihydrochloride combined with PD-1 antibody in patients with metastatic pancreatic cancer who failed to standard treatment.

DETAILED DESCRIPTION:
There is no standard treatment for patients with metastatic pancreatic cancer who failed to FOLFIRINOX or AG (consisting of Gemcitabine and Abraxane). Patients with metastatic pancreatic cancer who are unable to tolerate or have failed to respond to standard chemotherapy will be enrolled in this clinical trial. They will be administered a combination treatment of Sapropterin Dihydrochloride and PD-1 antibody. The primary endpoints of this study are objective response rate and safety. The secondary endpoints will encompass overall survival, progression-free survival, and quality of life. The study aims to enroll a total of 20 participants.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) confirmed pancreatic ductal adenocarcinoma (PDAC).
* Recurrent disease or metastatic disease evaluated by abdominal contrast-enhanced CT, MRI, and chest CT. PET/CT or other imaging examinations would be used if necessary.
* Fail or could not tolerate standard chemotherapy.
* ECOG score 0 or 1.
* Have measurable target lesion.
* Serum total bilirubin level is less than 1.5 x ULN. ALT and AST are less than 2 x ULN. Hemoglobin≥9g/dL, platelet≥75×10*9/L, white blood count ≥3.0×10*9/L, neutrophil ≥1.5×10*9/L. Serum creatinine ≤ 1.5 × ULN or creatinine clearance rate > 60 mL/min.
* Signed informed consent.

Exclusion Criteria:

* History of participation of other clinical trials within 4 weeks
* Known or suspected allergy to Sintilimab or tetrahydrobiopterin.
* Female patients during pregnancy or lactation.
* Patients who lack the ability to provide informed consent due to psychological, family, social, or other factors.
* Patients with a history of other malignant tumors besides pancreatic cancer before enrollment, except for non-melanoma skin cancer, carcinoma in situ of the cervix, or cured early-stage prostate cancer.
* Patients with severe cardiac, pulmonary, hepatic, or renal dysfunction, hematopoietic system diseases, cachexia, or other conditions that are intolerable to radiotherapy, chemotherapy, or surgery.
* Patients with autoimmune diseases, a history of autoimmune diseases (such as colitis, hepatitis, hyperthyroidism, including but not limited to these diseases or syndromes), as well as a history of immune deficiency, including HIV-positive test results, or other acquired or congenital immune deficiency diseases, or a history of organ transplantation and allogeneic bone marrow transplantation.
* Patients who require systemic corticosteroid therapy (> 10 mg/day prednisone equivalent dose) or other immunosuppressive drugs within 14 days before the first administration or during the study. However, the following situations are allowed for enrollment: In the absence of active autoimmune diseases, patients are allowed to use topical or inhaled steroids, or adrenal hormone replacement therapy at a dose ≤ 10 mg/day prednisone equivalent dose.
* Patients with a history of interstitial lung disease or non-infectious pneumonia.
* Patients with active pulmonary tuberculosis infection detected through medical history or CT examination, or a history of active pulmonary tuberculosis infection within 1 year before enrollment, or patients with a history of active pulmonary tuberculosis infection more than 1 year ago but without proper treatment.
* Subjects with active hepatitis B (HBV DNA ≥ 2000 IU/mL or 10*4 copies/mL), hepatitis C (positive hepatitis C antibody and HCV-RNA higher than the lower limit of detection of the analytical method).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Every 6 weeks (2 cycles) from first treatment to disease progression or totally 2 years Based on irRECIST
  The percentage of patients whose cancer shrinks or disappears after treatment
Adverse events by NCI-CTCAE v5.0 | Every 3 weeks from first treatment to disease progression or totally 2 years Based on irRECIST
  Safety and tolerability

SECONDARY OUTCOMES:
Overall Survival (OS) | up to approximately 2 year
  The time from registration to death due to any cause, or censored at date last known alive.
Progression-Free Survival (PFS) | up to approximately 1 year
  PFS as measured in accordance with the irRECIST version 1.1
EORTC QLQ-C30 survey | up to approximately 2 year
  Quality of life survey
EORTC-QLQ-PAN26 survey | up to approximately 2 year
  Quality of life survey

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer center of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No